CLINICAL TRIAL: NCT06252740
Title: Investigation of Regional Interdependence of the Hip and Spine in Baseball Players With Low Back Pain
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: A-ER-110-579
Record Dates: First submitted 2023-05-16; First posted 2024-02-12 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2023-11

CONDITIONS: Low Back Pain; Thoracic
Keywords: Baseball batting; Motion analysis; Regional interdependence,; Hip; Joint mobility; Muscle stiffness
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- control group: Baseball players without a history of low back pain
  Interventions: Other: No intervention
- experimental group: Baseball players with a history of low back pain
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Comare the difference in batting mechanics, hip and thoracic spine mobility, and muscle stiffness in baseball players with and without a history of low back pain

SUMMARY:
Low back pain (LBP) is a common musculoskeletal symptom in athletes. More than 40% percent of high school baseball players reported incidents of LBP during the previous year. University baseball athletes were 3.23 times more likely to have lumbar intervertebral disk degeneration than the nonathletic university students. According to the regional interdependence model, a patient's chief complaints may be directly or indirectly related to or influenced by physical impairments from various body systems and regardless of proximity to the primary symptom(s). Athletes with a chief complaint of LBP frequently demonstrate with mobility restrictions in the thoracic spine and hips, which may contribute to compensatory hypermobility in the lumbar spine and subsequently lead to LBP. Few studies have examined the relationship between thoracic spine mobility and LBP, while many studies investigating the relationship between hip joint mobility and LBP in athletes showed inconsistent results. The inconsistent results may be due to different types of sports and measurement methods. Therefore, the objectives of this research project are to: (1) examine if baseball players with a history of LBP have mobility restriction in the thoracic spine and hips and movement coordination within the spine and hip regions during baseball batting that are different from those without a history of LBP; (2) identify thoracic spine and hip joint mobility and coordination related predictors for batting velocity and LBP in baseball players. This 2-year research project plans to recruitment a total of 110 male baseball players aged between 18 and 30 years from university and community recreational league baseball teams (55 players with a history of LBP and 55 age-matched players without a history of LBP). Participants will receive physical examination for the thoracic spine and hip joints (joint mobility and muscle stiffness) and 3D motion analysis for baseball batting. The results of this research project will guide the development of more specific and effective treatment and preventative training for baseball players with LBP and enhance their batting performance.

ELIGIBILITY:
Inclusion Criteria:

• Baseball players who had experienced at least 2 episodes of LBP that limits their performance for a period of greater than 3 days in the previous year.

Exclusion Criteria:

* Current LBP symptoms including weakness and numbness in the lower extremities
* Previous surgery to the back, upper or lower extremities
* Marked spinal deformity (e.g., scoliosis, or kyphosis)
* Any other orthopedic or medical problem that would have limited their ability to fully participate in baseball training and competition in the last year.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: university and recreational leagues baseball teams
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-11-02 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Angular displacement of spine during baseball batting | immediately after enrollment
  Measured by the Vicon motion analysis system in the horizontal plane
Angular displacement of hip during baseball batting | immediately after enrollment
  Measured by the Vicon motion analysis system in the horizontal plane
Angular velocity of spine during baseball batting | immediately after enrollment
  Measured by the Vicon motion analysis system in the horizontal plane
Angular velocity of hip during baseball batting | immediately after enrollment
  Measured by the Vicon motion analysis system in the horizontal plane
Thoracic spine mobility | immediately after enrollment
  Measured by the Vicon motion analysis system in sitting

SECONDARY OUTCOMES:
Hip joint mobility | immediately after enrollment
  Ranges of hip internal and external rotation measured by inclinometer in sitting
Stiffness of biceps femoris muscle | immediately after enrollment
  Measured by the hand-held MyotonPRO device in N/m
Stiffness of rectus femoris muscle | immediately after enrollment
  Measured by the hand-held MyotonPRO device in N/m
Stiffness of tensor fasciae latae muscle | immediately after enrollment
  Measured by the hand-held MyotonPRO device in N/m
Stiffness of glutues maximus muscle | immediately after enrollment
  Measured by the hand-held MyotonPRO device in N/m
Stiffness of thoracic erector spinae muscle | immediately after enrollment
  Measured by the hand-held MyotonPRO device in N/m
FABER's test | immediately after enrollment
  Measured as distance between knee and bed in cm
Straight leg raising test | immediately after enrollment
  Measured as hip flexion angle (with knee extended) in degree
Modified Thomas test | immediately after enrollment
  Measured as hip flexion angle (with knee flexed) in degree
Ober test | immediately after enrollment
  Measured as hip adduction angle in degree

CONTACTS AND LOCATIONS:
Locations (1):
- National Cheng Kung University, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No